CLINICAL TRIAL: NCT01783678
Title: A Phase 3, Open-label Study to Investigate the Efficacy and Safety of Sofosbuvir Plus Ribavirin in Chronic Genotype 1, 2, 3 and 4 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Co-infected Subjects
Brief Title: A Phase 3, Open-label Study to Investigate the Efficacy and Safety of Sofosbuvir Plus Ribavirin in Chronic Genotype 1, 2, 3 and 4 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Co-infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0124
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis C; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Genotype 2 treatment-naive (Experimental): Treatment-naive (TN) participants with HIV-1 and genotype 2 HCV coinfection will receive sofosbuvir plus RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- Genotype 2/3 treatment-experienced (Experimental): Treatment-experienced (TE) participants with HIV-1 and genotype 2 or 3 HCV co-infection will receive sofosbuvir plus RBV for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- Genotype 1/3/4 treatment-naive (Experimental): Treatment naive (TN) participants with HIV-1 and genotype 1, 3, or 4 HCV co-infection will receive sofosbuvir plus RBV for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This is an Open-label Phase 3 study in adults with chronic genotypes 1, 2, 3, and 4 HCV infection who are co-infected with HIV-1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with HIV-1 and chronic HCV genotype 1, 2, 3, or 4 co-infection
* HCV RNA > 10,000 IU/mL at screening
* HCV treatment history:

  * Treatment-naive for HCV genotypes 1, 2, 3, or 4, or
  * Treatment-experienced for HCV genotypes 2 or 3
* HIV antiretroviral (ARV) criteria:

  * On a stable, protocol-approved, HIV ARV regimen with undetectable HIV RNA for > 8 weeks prior to screening, or
  * ARV untreated for ≥ 8 weeks prior to screening, with a CD4 T-cell count > 500 cells/mm^3
* Presence or absence of cirrhosis; a liver biopsy may be required
* Healthy according to medical history and physical examination with the exception of HCV and HIV diagnosis
* Agree to use two forms of highly effective contraception for the duration of the study and 6 months after the last dose of study medication

Exclusion Criteria:

* HCV genotype 1 or 4 with previous HCV treatment
* Poor control with HIV ARV regimen requiring a possible dose modification of therapy within 4 weeks of study medication dosing
* A new AIDS-defining condition diagnosed within 30 days prior to screening
* Prior use of any other inhibitor of the HCV NS5B polymerase
* History of any other clinically significant chronic liver disease
* Evidence of or history of decompensated liver disease
* Chronic hepatitis B virus (HBV) infection
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of immunosuppressive agents or immunomodulatory agents
* Clinically relevant drug or alcohol abuse within 12 months of screening
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the participant's participation for the full duration of the study or not be in the best interest of the participant in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Gaggar, MD, PhD, Study Director — Gilead Sciences
Locations (24):
- Australia (4):
  - Darlinghurst, New South Wales
  - Sydney, New South Wales
  - Melbourne, Victoria
  - Parkville, Victoria
- France (3):
  - Lyon
  - Nice
  - Paris
- Germany (6):
  - Berlin
  - Bonn
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Würzburg
- Italy (5):
  - Bergamo
  - Milan
  - Napoli
  - Rome
  - Torino
- Spain (3):
  - Barcelona
  - Madrid
  - Seville
- United Kingdom (3):
  - Glasgow
  - London
  - Sussex

REFERENCES:
- [Derived] Molina JM, Orkin C, Iser DM, Zamora FX, Nelson M, Stephan C, Massetto B, Gaggar A, Ni L, Svarovskaia E, Brainard D, Subramanian GM, McHutchison JG, Puoti M, Rockstroh JK; PHOTON-2 study team. Sofosbuvir plus ribavirin for treatment of hepatitis C virus in patients co-infected with HIV (PHOTON-2): a multicentre, open-label, non-randomised, phase 3 study. Lancet. 2015 Mar 21;385(9973):1098-106. doi: 10.1016/S0140-6736(14)62483-1. Epub 2015 Feb 4. PMID 25659285
- [Derived] Younossi ZM, Stepanova M, Sulkowski M, Naggie S, Puoti M, Orkin C, Hunt SL. Sofosbuvir and Ribavirin for Treatment of Chronic Hepatitis C in Patients Coinfected With Hepatitis C Virus and HIV: The Impact on Patient-Reported Outcomes. J Infect Dis. 2015 Aug 1;212(3):367-77. doi: 10.1093/infdis/jiv005. Epub 2015 Jan 12. PMID 25583164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 39 study sites in Australia and Europe. The first participant was screened on 18 January 2013. The last study visit occurred on 10 July 2014.
Pre-assignment Details: 346 participants were screened.
Groups:
- Genotype 2 Treatment-naive: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 12 weeks in treatment-naive participants with HIV-1 and genotype 2 HCV coinfection
- Genotype 1 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 1 HCV coinfection
- Genotype 2 Treatment-experienced: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-experienced participants with HIV-1 and genotype 2 HCV coinfection
- Genotype 3 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 3 HCV coinfection
- Genotype 3 Treatment-experienced: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-experienced participants with HIV-1 and genotype 3 HCV coinfection
- Genotype 4 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 4 HCV coinfection
Period: Overall Study
Arm/Group | Genotype 2 Treatment-naive | Genotype 1 Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Started | 19 | 112 | 6 | 58 | 49 | 31
Completed | 17 | 94 | 5 | 50 | 42 | 26
Not Completed | 2 | 18 | 1 | 8 | 7 | 5
Not completed — Randomized but Not Treated | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 13 | 1 | 3 | 6 | 5
Not completed — Lost to Follow-up | 0 | 4 | 0 | 2 | 1 | 0
Not completed — Withdrew Consent | 1 | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- Genotype 2 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks in treatment-naive participants with HIV-1 and genotype 2 HCV coinfection
- Total: Total of all reporting groups
Arm/Group | Genotype 2 Treatment-naive | Genotype 1 Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive | Total
Number analyzed (Participants) | 19 | 112 | 6 | 57 | 49 | 31 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8.2) | 45 (7.6) | 55 (10.2) | 47 (5.4) | 49 (6.2) | 47 (5.9) | 47 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 0 | 19 | 11 | 7 | 53
  Male | 15 | 100 | 6 | 38 | 38 | 24 | 221
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 3
  White | 18 | 104 | 5 | 54 | 49 | 29 | 259
  Asian | 0 | 5 | 0 | 2 | 0 | 0 | 7
  American Indian/Alaska Native/First Nations | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Not Permitted | 0 | 1 | 0 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 4 | 0 | 3 | 5 | 1 | 16
  Not Hispanic or Latino | 16 | 106 | 6 | 54 | 44 | 29 | 255
  Not Permitted | 0 | 2 | 0 | 0 | 0 | 1 | 3
Cirrhosis Status [Number; unit: participants]
  No | 18 | 95 | 4 | 54 | 26 | 23 | 220
  Yes | 1 | 17 | 2 | 3 | 23 | 8 | 54
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 12 | 48 | 3 | 30 | 25 | 9 | 127
    CT | 5 | 45 | 1 | 21 | 20 | 14 | 106
    TT | 2 | 18 | 2 | 6 | 4 | 8 | 40
    Missing | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.7 (0.66) | 6.3 (0.72) | 6.4 (0.62) | 6.3 (0.71) | 6.3 (0.77) | 5.9 (0.85) | 6.3 (0.75)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 2 | 33 | 1 | 21 | 12 | 12 | 81
  ≥ 6 log10 IU/mL | 17 | 79 | 5 | 36 | 37 | 19 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ, ie, < 25 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug. 1 participant with genotype 1 HCV infection did not have subtype information available.
Measure: Number; unit: percentage of participants
Groups:
- All Genotype 1 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 1 HCV coinfection
- Genotype 1a Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 1a HCV coinfection (subset of All Genotype 1 Treatment-naive reporting group)
- Genotype 1b Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 1b HCV coinfection (subset of All Genotype 1 Treatment-naive reporting group)
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 112 | 100 | 11 | 6 | 57 | 49 | 31
percentage of participants | 89.5 | 84.8 | 84.0 | 90.9 | 83.3 | 91.2 | 85.7 | 83.9

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants permanently discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- Genotype 2/3 Treatment-experienced: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-experienced participants with HIV-1 and genotype 2 or 3 HCV coinfection
- Genotype 1/3/4 Treatment-naive: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks in treatment-naive participants with HIV-1 and genotype 1, 3, or 4 HCV coinfection
Arm/Group | Genotype 2 Treatment-naive | Genotype 2/3 Treatment-experienced | Genotype 1/3/4 Treatment-naive
Number analyzed (Participants) | 19 | 55 | 200
percentage of participants | 0 | 1.8 | 3.5

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < the lower limit of quantitation (LLOQ) 4 weeks and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set. 1 participant with genotype 1 HCV infection did not have subtype information available.
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 112 | 100 | 11 | 6 | 57 | 48 | 31
percentage of participants
  SVR4 | 89.5 | 87.5 | 87.0 | 90.9 | 83.3 | 91.2 | 87.8 | 90.3
  SVR24 | 89.5 | 83.0 | 82.0 | 90.9 | 83.3 | 91.2 | 83.7 | 80.6

4. Secondary Outcome: HCV RNA Change From Baseline at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed. 1 participant with genotype 1 HCV infection did not have subtype information available.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 112 | 100 | 11 | 6 | 54 | 48 | 31
log10 IU/mL | -4.72 (0.573) | -4.54 (0.776) | -4.57 (0.777) | -4.35 (0.752) | -4.34 (0.575) | -4.41 (0.498) | -4.33 (0.667) | -4.21 (0.665)

5. Secondary Outcome: HCV RNA Change From Baseline at Week 2
Time Frame: Baseline; Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 111 | 99 | 11 | 6 | 55 | 47 | 30
log10 IU/mL | -5.29 (0.681) | -4.92 (0.717) | -4.97 (0.674) | -4.55 (0.928) | -4.98 (0.633) | -4.86 (0.677) | -4.89 (0.776) | -4.52 (0.843)

6. Secondary Outcome: HCV RNA Change From Baseline at Week 4
Time Frame: Baseline; Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 109 | 97 | 11 | 6 | 57 | 49 | 31
log10 IU/mL | -5.33 (0.655) | -4.95 (0.720) | -5.01 (0.674) | -4.55 (0.928) | -5.05 (0.618) | -4.89 (0.708) | -4.84 (0.895) | -4.57 (0.846)

7. Secondary Outcome: HCV RNA Change From Baseline at Week 6
Time Frame: Baseline; Week 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 109 | 97 | 11 | 6 | 57 | 49 | 31
log10 IU/mL | -5.33 (0.655) | -4.95 (0.718) | -5.01 (0.672) | -4.55 (0.928) | -5.05 (0.618) | -4.89 (0.710) | -4.91 (0.789) | -4.57 (0.846)

8. Secondary Outcome: HCV RNA Change From Baseline at Week 8
Time Frame: Baseline; Week 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 109 | 97 | 11 | 6 | 56 | 49 | 31
log10 IU/mL | -5.33 (0.655) | -4.95 (0.722) | -5.01 (0.676) | -4.55 (0.928) | -5.05 (0.618) | -4.88 (0.708) | -4.86 (0.876) | -4.57 (0.846)

9. Secondary Outcome: Percentage of Participants Experiencing Virologic Failure
Description: On-treatment virologic failure was defined as either:
  * Virologic breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Nonresponse (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment).
  Virologic relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period, having achieved HCV RNA < LLOQ at last on-treatment visit."
Time Frame: Baseline up to Posttreatment Week 24
Population: Full Analysis Set. 1 participant with genotype 1 HCV infection did not have subtype information available.
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 2 Treatment-naive | All Genotype 1 Treatment-naive | Genotype 1a Treatment-naive | Genotype 1b Treatment-naive | Genotype 2 Treatment-experienced | Genotype 3 Treatment-naive | Genotype 3 Treatment-experienced | Genotype 4 Treatment-naive
Number analyzed (Participants) | 19 | 112 | 100 | 11 | 6 | 57 | 49 | 31
percentage of participants
  On-Treatment Virologic Failure | 0 | 0 | 0 | 0 | 0 | 0 | 2.0 | 0
  Virologic Relapse | 5.3 | 12.5 | 13.0 | 9.1 | 16.7 | 7.0 | 12.5 | 16.1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Arm/Group | Genotype 2 Treatment-naive | Genotype 2/3 Treatment-experienced | Genotype 1/3/4 Treatment-naive
Serious Adverse Events (participants affected / at risk) | 0/19 | 5/55 | 10/200
Other Adverse Events (participants affected / at risk) | 17/19 | 45/55 | 166/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 2 Treatment-naive (N=19) | Genotype 2/3 Treatment-experienced (N=55) | Genotype 1/3/4 Treatment-naive (N=200)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Genotype 2 Treatment-naive (N=19) | Genotype 2/3 Treatment-experienced (N=55) | Genotype 1/3/4 Treatment-naive (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 16
Tachycardia (Cardiac disorders) | 1 | 2 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 32
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 24
Vomiting (Gastrointestinal disorders) | 0 | 1 | 13
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 9
Constipation (Gastrointestinal disorders) | 0 | 0 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 10
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 11 | 40
Asthenia (General disorders) | 1 | 11 | 32
Pyrexia (General disorders) | 0 | 3 | 5
Influenza like illness (General disorders) | 1 | 0 | 4
Malaise (General disorders) | 1 | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 1 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 13
Rhinitis (Infections and infestations) | 1 | 0 | 8
Sinusitis (Infections and infestations) | 1 | 1 | 7
Bronchitis (Infections and infestations) | 1 | 0 | 7
Influenza (Infections and infestations) | 0 | 3 | 4
Pharyngitis (Infections and infestations) | 1 | 0 | 3
Ear infection (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urethritis gonococcal (Infections and infestations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 17
Hyperphagia (Metabolism and nutrition disorders) | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 11
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 7 | 35
Lethargy (Nervous system disorders) | 1 | 1 | 15
Dizziness (Nervous system disorders) | 0 | 5 | 9
Insomnia (Psychiatric disorders) | 3 | 5 | 36
Irritability (Psychiatric disorders) | 1 | 6 | 20
Anxiety (Psychiatric disorders) | 0 | 3 | 15
Sleep disorder (Psychiatric disorders) | 1 | 1 | 13
Depression (Psychiatric disorders) | 0 | 5 | 9
Depressed mood (Psychiatric disorders) | 2 | 0 | 4
Mood swings (Psychiatric disorders) | 1 | 1 | 2
Stress (Psychiatric disorders) | 1 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 11
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 16
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years